CLINICAL TRIAL: NCT02228200
Title: A Nurse-led Care Program on Quality of Life and Health Care Utilization for Cancer Patients in a Chemotherapy Day Center: A Randomized Controlled Trial
Brief Title: Nurse-led Care Program for Cancer Patients in Chemotherapy Day Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Shirley Siu Yin CHING, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: POLYU-HSEARS20120117002
Record Dates: First submitted 2014-08-19; First posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Breast Neoplasms; Colorectal Neoplasms
Keywords: Oncology Nursing; Advanced Practice Nursing; Nurse-led care; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse-led care (Experimental): Subjects in the nurse-led care arm received nurse-led care and routine care.
  Interventions: Behavioral: Nurse-led care; Behavioral: Routine care
- Routine care (Active Comparator): Subjects in the routine care arm received routine care provided by the study hospital.
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Nurse-led care — The nurse-led care consisted of a pre-chemotherapy nursing consultation and telephone follow-up sessions during chemotherapy. The nursing consultation was on the day of the first cycle before drug administration. It included: history review, overall status evaluation, need and problem assessment, information provision, psychological support, and referral. The telephone follow-up sessions were delivered within one week after the 1st, 2nd, 4th, and 6th, and 8th cycle. A telephone follow-up session included: (i) The overall status assessment and problem triage; (ii) Care delivery based on problem severity; (iii) Evaluation of the change of the problems on the following telephone call.
  Arms: Nurse-led care
Behavioral: Routine care — Routine care includes: (1) Brief education on possible side-effects and coping skills before chemotherapy; (2) Care on chemotherapy day: vital sign assessment, casual communication between nurses and patients, video about chemotherapy and side effects management. (3) Care in chemotherapy intervals: hotline for patients when they have health problems at home.

SUMMARY:
A nurse-led care program for cancer patients receiving chemotherapy in an outpatient setting was formulated. The aim of the study was to assess the effect of this nurse-led care program on cancer patients who received neo-adjuvant/adjuvant chemotherapy in a chemotherapy day center in terms of quality of life, symptom experiences, self-efficacy, health care utilization, and satisfaction with care. Specifically, the objectives are:

* To compare the differences of health care utilization between the two arms.
* To compare the differences of cancer patients' satisfaction with care between the two arms.
* To explore the experiences of cancer patients in the intervention arm.
* To understand the experiences of the intervention nurses of the program and their opinions on further development.

DETAILED DESCRIPTION:
Chemotherapy affects cancer patients in many ways. It is common that patients suffer multiple side-effects simultaneously. Psychological distress is also a common problem during chemotherapy. Distressful experiences in chemotherapy may lead to deterioration in a patient's of quality of life (QOL). In addition, cancer patients have particularly high unmet needs during treatment, including informational needs, psychosocial needs, needs in the activities of daily living, supportive care needs, sexual needs, and communication needs. Among them, information is the most frequently reported need in the treatment phase. These unmet needs cause uncertainty, anxiety, and distress to cancer patients.

Outpatient-based chemotherapy is now widely established. Despite its benefits to health care institutions and cancer patients, there are attendant challenges. Cancer patients need to take care of themselves at home during each interval of chemotherapy. Without adequate support from health care providers, cancer patients may not be able to properly manage chemotherapy and its effects by themselves. The poor management of side-effects may lead to increased health care utilization. Cancer patients need to develop new self-care skills to cope with chemotherapy.

Facing increasing numbers of cancer patients and burgeoning health care needs, health care professionals must address the issue of how to improve the quality of care during chemotherapy. Nurse-led care is a highly recommended and innovative way of improving quality of care. It shows distinct advantages in terms of providing holistic care because it is based on the philosophy of the uniqueness of individuals and the multidimensionality of human beings. The feasibility and effects of nurse-led care are being explored in an increasing number of studies. However, studies of nurse-led care for cancer patients receiving outpatient-based chemotherapy are far away adequacy. There is a need to examine the feasibility and effects of nurse-led care for cancer patients receiving chemotherapy in outpatient settings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary breast /lung/stomach/colorectal cancer;
* Receive chemotherapy for the first time;
* Karnofsky performance scale equal or over 60;
* Communicate with Cantonese and read Chinese;
* Can be contacted with telephone.

Exclusion Criteria:

* Having a history of psychiatric or intellectual impairment such as: dementia, schizophrenia, mental retardation, depression, and anxiety disorder;
* Having received CT before either in the study hospital or other hospital;
* Receive concurrent chemoradiotherapy;
* At the end stage of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | T0: before chemotherapy (week 0); T1: in the middle of chemotherapy (i.e. week 4 to 10); T2: three weeks after last cycle of chemotherapy (i.e. week 13 to 20).
  Questionnaire: Quality of life will be assessed by the Chinese version of the Functional Assessment of Cancer Therapy-General Scale (FACT-G)

SECONDARY OUTCOMES:
Health care utilization | During chemotherapy (i.e. from week 0 to week 20)
  Five types of health care service will be collected: patient-initiated telephone calls, clinical visits to oncology outpatient department, clinical admission (from oncology outpatient department), emergency room visits, and hospital admission (from emergency room).

OTHER OUTCOMES:
Change in Symptom prevalence and distress levels | T0: before chemotherapy (i.e. week 0); T1: in the middle of chemotherapy (week 4 to 10); T2: three weeks after last cycle of chemotherapy (i.e. week 13 to 20).
  Questionnaire: The prevalence rates and distress levels caused by chemotherapy-related symptoms will be assessed by the Chemotherapy Symptom Assessment Scale (CSAS).
Satisfaction with care | At the end of chemotherapy (i.e. week 13 to 20)
  Satisfaction with care is evaluated by self-designed questionnaires.
Change in Self-efficacy | T0: before chemotherapy (week 0); T1: in the middle of chemotherapy (week 4 to 10); T2: three weeks after last cycle of chemotherapy (weel 13 to 20).
  Questionnaire: Self-efficacy will be assessed by the Strategies Used by People to Promote Health (SUPPH).
Subjects' experience | Three weeks after the last cycle of chemotherapy (i.e. week 13 to 20)
  Individual interviews will be adopted to understand the subjects' experiences, level of satisfaction, comments on further improvement of the care.
Intervention nurses' experience | At the end of data collection (week 20)
  Intervention nurses will be interviewed individually to understand their experiences of involving in the study and their comments on further improvement of the care.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Siu Yin CHING, PHD, Principal Investigator — School of Nursing, the Hong Kong Polytechnic Universtiy
Locations (1):
- Department of Clinical Oncology, Queen Elizabeth Hospital, Hong Kong, China

REFERENCES:
- [Derived] Lai XB, Ching SSY, Wong FKY, Leung CWY, Lee LH, Wong JSY, Lo YF. A Nurse-Led Care Program for Breast Cancer Patients in a Chemotherapy Day Center: A Randomized Controlled Trial. Cancer Nurs. 2019 Jan/Feb;42(1):20-34. doi: 10.1097/NCC.0000000000000539. PMID 28926349